CLINICAL TRIAL: NCT02708108
Title: Improving Diet and Exercise in Acute Lymphoblastic Leukemia (IDEAL Weight in ALL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Gabrielle's Angel Foundation (Other)
Responsible Party: Principal Investigator, Etan Orgel, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-14-00073
Record Dates: First submitted 2016-03-07; First posted 2016-03-15 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: B Precursor Type Acute Leukemia
MeSH Terms: interventions — Diet Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obesity Intervention (Experimental): Personalized 28-day Dietary Intervention and Activity and Exercise Intervention with the goal to reduce fat gain and lean muscle loss while inducing an overall negative energy balance.
  Interventions: Behavioral: Dietary Intervention; Behavioral: Activity and Exercise Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — Beginning at time of diagnosis, the dietary component of the intervention uses a personalized menu to implement high protein, moderate fat, and low glycemic index/high fiber diet to achieve a minimum net -10% daily caloric deficit during the induction phase of chemotherapy.
Behavioral: Activity and Exercise Intervention — Beginning at the time of diagnosis, the exercise and activity component uses an "activity menu" to implement a target level of 200 minutes per week of moderate exercise activity (as estimated by metabolic equivalents) during the induction phase of chemotherapy.

SUMMARY:
This study tests the ability of a focused dietary, exercise, and activity intervention to reduce fat gain during induction therapy for childhood acute lymphoblastic leukemia to improve disease response and reduce toxicity.

DETAILED DESCRIPTION:
In our previous study, we have observed that: 1) nearly half ALL patients are overweight or obese at diagnosis, 2) all patients, regardless of starting weight, gain significant fat mass over the first month of therapy (on average 20-30%), and 3) obesity at the time of diagnosis is associated with a higher likelihood of poor response to chemotherapy as evidenced by persistent leukemia (minimal residual disease) after induction therapy. Together, these data show that body fat is a significant risk factor for ALL treatment failure, and that its negative effects are evident within the first month of treatment. Recent laboratory and clinical data illustrates the ability of diet restriction and physical activity to improve chemotherapy efficacy, reduce treatment-related toxicities and better overall quality of life.

Given the importance of successful induction therapy for ALL in predicting long term survival and the negative role of obesity on treatment success, this study tests a complete personalized dietary and exercise intervention for pre-adolescents, adolescents, and young adults newly diagnosed with B-precursor ALL ("pre-B ALL") that aims to reduce fat gained during induction therapy and thereby improve treatment response, toxicity rates, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 10 years of age and less than or equal to 21 years of age at time of diagnosis
* Have a new diagnosis of untreated NCI/Rome High Risk B-precursor ALL (HR-ALL)
* Are beginning treatment on- or as per- a Children's Cancer Group/Children's Oncology Group (CCG-COG) protocol with a 4-drug Induction including vincristine, daunorubicin (or doxorubicin), asparaginase, and at least 14 days of glucocorticoid steroids

Exclusion Criteria:

* Have a diagnosis of Down syndrome (Trisomy 21) or any genetic disease associated with abnormal body composition
* Be underweight or "at risk for underweight" with moderate weight loss, defined as a starting Body Mass Index (BMI) <10th percentile for age and sex (for those >20 years of age, defined as an absolute BMI < 18.5)
* Have pre-existing abnormal intestinal function (e.g. protein-wasting enteropathy, fat malabsorption)
* Be unable to comply with the recommended diet or activity interventions (as determined by study or treatment team)
* Have a history of prior chemotherapy or radiation for other cancers
* Be unable to complete the necessary radiology examinations with fully interpretable data (e.g. hip replacement and metal prostheses preclude evaluation by DXA)
* Be pregnant (to be confirmed by urine or serum pregnancy test as per institutional routine care for chemotherapy and radiology exams)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2019-04 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etan Orgel, MD MS, Principal Investigator — Children's Hospital Los Angeles; Steven D Mittelman, MD PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orgel E, Framson C, Buxton R, Kim J, Li G, Tucci J, Freyer DR, Sun W, Oberley MJ, Dieli-Conwright C, Mittelman SD. Caloric and nutrient restriction to augment chemotherapy efficacy for acute lymphoblastic leukemia: the IDEAL trial. Blood Adv. 2021 Apr 13;5(7):1853-1861. doi: 10.1182/bloodadvances.2020004018. PMID 33792627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A non-prospective, historical cohort was used as a comparison group for this single-arm study.
Groups:
- Obesity Intervention: Diet: 10% caloric deficit, protein >= 20% calories, fat <25% calories, carbohydrate <55% calories, low glycemic load <100/2000 kcal.
  Activity: 200 minutes/week of aerobic and resistance training
  Duration 28 days
- Historical Control: Previous, consecutively treated unselected patients with B-ALL without the IDEAL intervention
Period: Overall Study
Arm/Group | Obesity Intervention | Historical Control
Started | 40 | 83
Completed | 38 | 80
Not Completed | 2 | 3
Not completed — Death | 1 | 2
Not completed — Regimen change | 1 | 0
Not completed — No MRD and no imaging available | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Historical Control: Historical control assembled from previous, unselected, consecutive patients treated for B-ALL matching eligibility criteria.
- Total: Total of all reporting groups
Arm/Group | Obesity Intervention | Historical Control | Total
Number analyzed (Participants) | 40 | 80 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (3.0) | 14.7 (2.5) | 14.80 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 37 | 53
  Male | 24 | 43 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 66 | 92
  Not Hispanic or Latino | 8 | 14 | 22
  Unknown or Not Reported | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 40 | 80 | 120
BMI Category [Count of Participants; unit: Participants] — BMI category assigned as per Center for Disease Control & Prevention age and sex normalized values for ages <20 years of age (Absolute BMI for age 20 years and older).
  Lean BMI%ile 10 to 84.9 (BMI 18.5 to <25) Overweight BMI%ile 85-94.9 (BMI 25-29) Obese BMI%ile >=95 (BMI >=30)
  Participants
    Lean | 14 | 45 | 59
    Overweight | 6 | 9 | 15
    Obese | 20 | 26 | 46

OUTCOME MEASURES:

1. Primary Outcome: Fat Mass
Description: Assessment of change in fat before and after the induction chemotherapy phase (first 28 days of chemotherapy) as measured dual-energy x-ray absorptiometry (DXA) in comparison to fat gain in a recent historical cohort. Calculated as (Day 28 Fat Mass - Diagnosis Fat Mass)/Diagnosis Fat Mass
Time Frame: Diagnosis and 28-35 days
Population: Includes enrolled (or from historical control) with imaging information via DXA scan.
Measure: Median (Inter-Quartile Range); unit: percent change in fat mass
Arm/Group | Obesity Intervention | Historical Control
Number analyzed (Participants) | 36 | 36
percent change in fat mass | 5.1 [-0.70 to 15.13] | 10.7 [3.29 to 19.28]

2. Secondary Outcome: Percentage of Participants With Minimal Residual Disease >=0.01%
Description: Compare the rate of minimal residual disease "positivity" (defined as >=0.01%) in the bone marrow by flow cytometry after the induction phase of chemotherapy as compared to a recent historical cohort
Time Frame: 28-35 days from diagnosis
Measure: Count of Participants; unit: Participants
Groups:
- Historical Control: Previous, consecutively treated unselected patients with B-ALL
Arm/Group | Obesity Intervention | Historical Control
Number analyzed (Participants) | 38 | 80
Participants | 12 | 30
Statistical Analysis 1: Comparison: Obesity Intervention vs Historical Control; Test type: Other — Multivariable analysis; p = 0.02, Regression, Logistic — Reported as 1-sided p-value; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.09 to 0.92] — Multivariable model includes age, BMI category, cytogenetic risk, ethnicity, sex

3. Secondary Outcome: Percentage of Successfully Completed Visits With Study Dietitian and Study Physiotherapist
Description: Assess feasibility of incorporating the intervention into induction chemotherapy as defined by >80% of overall scheduled study visits successfully completed. The expected number of overall visits is equal to the sum of total visits scheduled with the physiotherapist (PT) or the registered dietitian (RD). The measure was calculated as the total # expected visits/completed visits.
Time Frame: 28 days
Population: A total of 392 visits with the PT or RD were expected to be completed as part of the the study intervention.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Obesity Intervention
Number analyzed (Participants) | 40
Number analyzed (Visits) | 392
Visits | 339

4. Secondary Outcome: Percentage of Overall Adherence to the IDEAL Intervention
Description: Overall adherence to the study intervention was calculated as the mean of dietary adherence (average of percent consumed calories/prescribed calories for each food group) and activity (self-reported % adherence to prescribed days).
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: % adherence
Arm/Group | Obesity Intervention
Number analyzed (Participants) | 39
% adherence | 82.1 [77.7 to 86.5]

ADVERSE EVENTS:
Time Frame: A maximum of 35 days from enrollment (i.e., Induction phase only)
Description: Adverse event (AE) reporting was targeted and included: nil per os (NPO, 'nothing by mouth') due to toxicity, use of naso-gastrointestinal/nasojejunal (NG/NJ) or parenteral nutrition, any surgeries, any ICU admissions, Grade 3 or 4 hepatic or pancreatic toxicity, presence of osteonecrosis or fracture. Toxicities due to underlying chemotherapy were not attributable to the intervention and were not captured.
  AE data was unavailable for the historical cohort.
Groups:
- Historical Control: Historical control group
  Prospective adverse event reporting is NOT available for this group. Zero reflected below therefore reflects the absence of prospective reporting in this arm.
Arm/Group | Obesity Intervention | Historical Control
All-Cause Mortality (participants affected / at risk) | 1/40 | 2/80
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/80
Other Adverse Events (participants affected / at risk) | 0/40 | 0/80

LIMITATIONS AND CAVEATS:
Adverse event reporting was not available from the historical cohort for comparison with the IDEAL cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT02708108/Prot_SAP_000.pdf